CLINICAL TRIAL: NCT04112485
Title: Open Discectomy Versus Microscope Assisted Discectomy for Treatment of Symptomatic Lumbar Disc Herniation: a Comparative Study
Brief Title: Open Discectomy Versus Microscopic Discectomy for Lumbar Disc Herniation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Sherwan Ahmed Ali Hamawandi, assistant professor of orthopedic surgery, Hawler Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMU/Sherwan3
Record Dates: First submitted 2019-09-27; First posted 2019-10-02 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Lumbar Disc Herniation
Keywords: Lumbar disc herniation , Open Discectomy, Micrdiscectomy
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open discectomy (Other): This group of patients are treated by open discectomy
  Interventions: Procedure: Microdiscectomy
- Microdiscectomy (Other): This group of patients are treated by Microdiscectomy
  Interventions: Procedure: Microdiscectomy

INTERVENTIONS:
Procedure: Microdiscectomy
  Other Names: Open discectomy

SUMMARY:
60 patients involved were divided into two matched groups; Group A: 30 patients were treated with conventional fenestration laminectomy and discectomy and Group B: 30 patients were treated with microdiscectomy. The age of the patients involved in this study ranged from 19 years old to 46 years old

DETAILED DESCRIPTION:
60 patients involved were divided into two matched groups; Group A: 30 patients were treated with conventional fenestration laminectomy and discectomy and Group B: 30 patients were treated with microdiscectomy. The age of the patients involved in this study ranged from 19 years old to 46 years old. All the patient was suffering from symptomatic lumbar disc herniation L4-5. Each patient was assessed clinically and MRI was done for all the patients to prove clinically, the symptomatic lumbar disc herniation which was present in all patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults who are symptomatic lumbar disc herniation L4-5. Each patient was assessed clinically and MRI was done for all the patients to prove clinically, the symptomatic lumbar disc herniation which was present in all patients. Conservative treatment for 6weeks was failed

Exclusion Criteria:

* smoking, previous lumbar spine surgery, Diabetes Melitus (DM) and neuromuscular disorders.

Ages: 19 Years to 46 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-03-04 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
Visual analogue score | Visua analogue score was assessed preoperatively and postoperatively to see how much change in pain can occurred after open discectomy and after Microdiscectomy for 1 year
  Visual analogue score of back pain and leg pain which represent a score from 0-10 so if patient has no pain so gives 0 and if has severe pain gives 10
Oswestry disability index | Oswestry disability index was assessed preoperatively and postoperatively to assess how much changes can occur after open discectomy and Microdiscectomy for 1 year after surgery
  Oswestry disability index in a measurement of functional ability of patients regarding pain and daily activities

REFERENCES:
- [Derived] Hamawandi SA, Sulaiman II, Al-Humairi AK. Open fenestration discectomy versus microscopic fenestration discectomy for lumbar disc herniation: a randomized controlled trial. BMC Musculoskelet Disord. 2020 Jun 15;21(1):384. doi: 10.1186/s12891-020-03396-x. PMID 32539752